CLINICAL TRIAL: NCT01830010
Title: A Two-part, Single- and Two Arm Randomized, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy (in Part 2 Only) of KRP203 in Patients Undergoing Stem Cell Transplant for Hematological Malignancies
Brief Title: A Two-part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of KRP203 in Patients Undergoing Stem Cell Transplant for Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CKRP203A2105
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2018-11

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Part 1: KRP203 (Experimental): All patients to receive KRP203 for 111days
  Interventions: Drug: Study Part 1: KRP203
- Study Part 2: lower KRP203 dose (Experimental): in this treatment arm patients will receive the lower KRP203 dose for 111 days on top of the standard treatment with cyclosporine A and methotrexte for GVHD prophylaxis
  Interventions: Drug: Study Part 2: KRP203 lower dose
- Study Part 2: higher KRP203 dose (Experimental): in this treatment arm patients will recieve the higher KRP203 dose for 111 days on top of standard treatment with tacrolimus and methotrexate for GVHD prophylaxis
  Interventions: Drug: Study Part 2: KRP203 higher dose

INTERVENTIONS:
Drug: Study Part 1: KRP203 — All subjects will receive KRP203 for 111 days
  Arms: Study Part 1: KRP203
Drug: Study Part 2: KRP203 lower dose
  Arms: Study Part 2: lower KRP203 dose
Drug: Study Part 2: KRP203 higher dose
  Arms: Study Part 2: higher KRP203 dose

SUMMARY:
Two part study to evaluate the safety, tolerability, pharmacokinetics, and efficacy (in Part 2 only) of KRP203 in patients undergoing allogeneic hemopoietic stem cell transplant for hematological malignancies

ELIGIBILITY:
Inclusion Criteria

* Patients aged 18 to 65 years, inclusive
* Patients must have a hematological malignancy that as per standard medical practice requires myeloablative conditioning (including short term myeloablative reduced intensity conditioning) followed by allogeneic hematopoetic stem cell transplant

  * Karnofsky Performance status ≥60%.
  * Suitable stem cell source available according to the graft selection algorithm using T-cell replete peripheral stem cells as a graft source

Exclusion Criteria:

* Resting heart rate below 55
* Significant cardiac disease (such as arrhytmia, heart failure) or any significant condition which in the investigators opinion would make the patient ineligible

  * Previous allogeneic HSCT
  * Any drug required that is not compatible with KRP203 (e.g. beta-blockers or anti-thymocyte globulin)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-06-28 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of safety | 111 days
  Safety and tolerability of KRP203 in patients undergoing allogeneic hematopoetic stem cell transplant for hematological malignancies

SECONDARY OUTCOMES:
Plasma Pharmacokinetics of KRP203: Area under the Plasma Concentration-time Curve (AUC) | 111 days
  The main PK parameters will be determined in whole blood using non-compartmental methods. Pk parameters being measured are: AUCtau AUC during a dosing interval (tau) of 24 hours [h.ng/mL] , AUCtauR Molar ratios between KRP203-P and KRP203 based on Cmax or AUCtau
Plasma Pharmacokinetics (PK) of KRP203: Observed Maximum Plasma Concentration Following Drug Administration (Cmax) | 111 days
  Cmax Maximum (peak) blood drug concentration after drug administration [ng/mL]
Plasma Pharmacokinetics (PK) of KRP203: Time to reach the maximum concentration after drug administration | 111 days
  Tmax Time to reach maximum (peak) concentration [ng/mL]
GVHD-free, relapse free survival | 1 years post-transplant
  occurence of GVHD, disease relaps and death will be assessed
GVHD-free, relapse free survival | 2 years post transplant
  occurence of GVHD, disease relaps and death will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Novartis Investigative Site, Paris, France
- Germany (5):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Jena
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Dertschnig S, Gergely P, Finke J, Schanz U, Holler E, Holtick U, Socie G, Medinger M, Passweg J, Teshima T, Stylianou C, Oehen S, Heim D, Bucher C. Mocravimod, a Selective Sphingosine-1-Phosphate Receptor Modulator, in Allogeneic Hematopoietic Stem Cell Transplantation for Malignancy. Transplant Cell Ther. 2023 Jan;29(1):41.e1-41.e9. doi: 10.1016/j.jtct.2022.10.029. Epub 2022 Nov 4. PMID 36343893
- See also: Results for CKRP203A2105 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17443
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=296